CLINICAL TRIAL: NCT01966848
Title: Comparison of Vanguard XP and Vanguard CR Total Knee Arthroplasties. A Randomized Controlled Trial Evaluating Early Component Migration by RSA and Patient Reported Outcome.
Brief Title: Comparison of Vanguard XP and Vanguard CR Total Knee Arthroplasties. A Trial Evaluating Early Component Migration by RSA and Patient Reported Outcome.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Principal Investigator, Morten Grove Thomsen, MD, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-1-2013-086
Record Dates: First submitted 2013-10-16; First posted 2013-10-22 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-11

CONDITIONS: Osteoarthritis
Keywords: Knee; osteoarthritis; arthroplasty; tka; rsa
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vanguard CR (Active Comparator): Patients will receive the posterior cruciate retaining Vanguard CR prosthesis
  Interventions: Device: Wich prosthesis is used
- Vanguard XP (Active Comparator): Patients will receive the bi-cruciate retaining Vanguard xp prosthesis
  Interventions: Device: Wich prosthesis is used

INTERVENTIONS:
Device: Wich prosthesis is used

SUMMARY:
In the history of TKA several different types of prosthetic designs have been evolved in order to optimize knee function after total knee replacement. The most common difference between the prosthetic designs revolves around issues concerning the preservation of the cruciate ligaments. The most popular prostheses have been the posterior stabilized prosthesis (PS) in which both cruciate ligaments are resected and the posterior cruciate retaining prosthesis (CR) in which only ACL is resected and PCL is preserved. Both these prosthetic designs have shown excellent clinical results in the literature.

In the knee the role of the cruciate ligaments is to insure anterior/posterior stability, but studies have also shown, that the cruciate ligaments contain proprioceptive mechanisms which control joint kinematics essential for accurate knee function. One could therefore imagine that a prosthetic design that preserves both cruciate ligaments would be superior to prosthetic designs in which ACL or ACL/PCL is resected in achieving good clinical results and patient satisfaction.

Only a few prosthetic designs, which preserve both cruciate ligaments, have been available to the market. However studies based on fluoroscopic assays and gait analysis has shown that this prosthetic design is superior to cruciate sacrificing designs in preserving normal knee kinematics during activities of daily living after TKA. Studies, in which patients have received two different types of prosthesis in each knee, have also shown that bi-cruciate retaining TKA's is preferred, when compared to more constrained prosthetic designs.

The new Vanguard XP TKA system (Biomet®, Warsaw, Indiana, USA) is a further development of the Vanguard TKA system, which has shown good clinical results in earlier studies. With the new Vanguard XP system both cruciate ligaments are preserved. In theory this should result in a more natural feeling of the knee because the stability and proprioceptive signals from both cruciate ligaments are preserved. In order to investigate the potential benefits of this new prosthetic design, the clinical and radiological results of knees receiving a Vanguard XP and Vanguard CR prostheses are compared.

In this study we wish to investigate:

1. If the use of the Vanguard XP prosthesis will influence the migration of the femur- and tibial components measured by Radiostereometric Analysis (RSA) when compared to the Vanguard CR prosthesis.
2. If the use of the Vanguard XP prosthesis will result in increased participant knee function, satisfaction and quality of life when compared to the Vanguard CR prosthesis.
3. If the use of the Vanguard XP prosthesis will influence radiologic signs of osteolysis, complication rates and revision rates when compared to the Vanguard CR prosthesis.

This project is carried out as a randomized controlled double-blinded trial, in which the clinical and radiological outcomes after treatment of knee osteoarthritis with insertion of either a Vanguard XP or Vanguard CR prosthesis is compared.

DETAILED DESCRIPTION:
1. Objectives Primary objective The primary objective of this study is to compare stability and fixation by RSA of Vanguard XP to that of Vanguard CR.

Secondary objective Secondary objective of this study is to assess the patient reported outcomes of Vanguard XP in comparison to Vanguard CR.

2. Background The primary goal of Total Knee Replacement surgery in the treatment of knee osteoarthritis is to reduce pain and restore knee function (stability and range of motion) in order to increase patient mobility and quality of life.

At Copenhagen University Hospital of Hvidovre, patients with severe osteoarthritis of the knee are treated with insertion of a cemented total knee prosthesis in which the anterior cruciate ligament is resected and the posterior cruciate ligament is retained (CR).

In the history of TKA several different types of prosthetic designs have been evolved in order to optimize knee function after total knee replacement. Most differences between the prosthetic designs revolve around issues concerning the preservation of the cruciate ligaments. The most popular prostheses used have been the posterior stabilized prosthesis (PS) in which both cruciate ligaments are resected and the posterior cruciate retaining prosthesis (CR) in which only ACL is resected and PCL is preserved. Both these prosthetic designs have shown excellent clinical results in the literature.

In the knee the role of the cruciate ligaments is to insure anterior/posterior stability, but studies have also shown, that the cruciate ligaments contain proprioceptive mechanisms which control joint kinematics essential for accurate knee function. One could therefore imagine that a prosthetic design that preserves both cruciate ligaments would be superior to prosthetic designs in which ACL or ACL/PCL is resected in achieving good clinical results and patient satisfaction.

Only a few prosthetic designs, which preserve both cruciate ligaments, have been available to the market. However studies based on fluoroscopic assays and gait analysis has shown that this prosthetic design is superior to cruciate sacrificing designs in preserving normal knee kinematics during activities of daily living after TKA13-16. Studies, in which patients have received two different types of prosthesis in each knee, have also shown that bi-cruciate retaining TKA's is preferred, when compared to more constrained prosthetic designs17-19.

The new Vanguard XP TKA system (Biomet®, Warsaw, Indiana, USA) is a further development of the Vanguard TKA system, which has shown good clinical results in earlier studies11-12. With the new Vanguard XP system both cruciate ligaments are preserved. In theory this should result in a more natural feeling of the knee because the stability and proprioceptive signals from both cruciate ligaments are preserved. In order to investigate the potential benefits of this new prosthetic design, the clinical and radiological results of knees receiving a Vanguard XP and Vanguard CR prostheses are compared.

In this study we wish to investigate:

1) If the use of the Vanguard XP prosthesis will influence the migration of the femur- and tibial components measured by Radiostereometric Analysis (RSA) when compared to the Vanguard CR prosthesis.

2) If the use of the Vanguard XP prosthesis will result in increased participant knee function, satisfaction and quality of life when compared to the Vanguard CR prosthesis.

3) If the use of the Vanguard XP prosthesis will influence radiologic signs of osteolysis, complication rates and revision rates when compared to the Vanguard CR prosthesis.

3. Device description Please see separate application for premarket testing. The Vanguard XP (with the XP tibial tray and XP tibial bearing to be used in this study) is not yet CE-marked.

4. Project design Project type This project is carried out as a randomized controlled double-blinded trial, in which the clinical and radiological outcomes after treatment of knee osteoarthritis with insertion of either a Vanguard XP or Vanguard CR prosthesis are compared.

After informed consent is obtained, participants are randomized to receive either a Vanguard XP or Vanguard CR prosthesis. Allocation of the patient to one of the two treatment groups is done in the operating room after surgical verification of both cruciate ligaments being intact. Non-transparent envelopes are used for the randomization process. Participants are unaware of which prosthesis they receive and the research coordinator handling the collected questionnaires postoperatively is also unaware of which prosthesis the patient has received.

Time schedule Recruitment of participants to this project is expected to begin in October 2013 or as soon as permission from the local Ethics Committee and the National Board of Health is obtained. 50 participants are to be randomized (25 participants in each study group). Recruitment is expected completed after a period of 1 year. Inclusion and randomization of approximately 5 participants per month is considered realistic regarding the logistical capacity for the additional necessary studies in this study. The project is expected to be completed 10 years after recruitment of the last participant (fall of 2024).

Participant termination At their own will participants can choose to leave the project at any time. Participants can also be withdrawn from the project at any time, if this is considered necessary by the investigators, e.g. in the event of deep infection leading to replacement of the prosthesis or long-term immobilisation because of comorbidity. If a participant is withdrawn or rescinds their consent, a "Lost to Follow-up" case report form will be completed detailing the reason for the participant's withdrawal.

Data recording Data relevant for this project will be registered in a data sheet. An individual data sheet will be kept for each recruited participant. Data will also be aggregated and stored electronically. The storage of data will be done according to the rules posted by the Danish Data Protection Agency. This project will be notified to and approved by the Danish Data Protection Agency before recruitment of partisipants is initiated.

5. Participant population 50 participants with knee osteoarthritis set to receive primary cemented total knee prosthesis at Copenhagen University Hospital Hvidovre.

Number of participants 50 recruited patients (25 in each group) are randomized to receive either Vanguard XP or Vanguard CR prosthesis.

Patients may be excluded intraoperatively, before randomization, if one or both of the cruciate ligaments are found to be missing or totally ruptured. We estimate that 20 % of enrolled patients will be excluded due to this, and therefore recruitement of 60 patients is needed.

Prior to recruitement of patients for the randomized study we will conduct a pilot study which will include 5 patients who will all receive the Vanguard XP.

The study's primary outcome measure is implant migration measured by RSA. If the minimally relevant total migration of the prosthesis measured by RSA is set to 0.2 mm1 then a total of 18 participants must be enrolled in each study group to show a statistically significant difference (95 % confidence, 80 % power).

In this study 2 x 25 participants are included. This will insure sufficient statistical power despite a dropout of 20%.

The power calculation is based on reaching sufficient power when a comparison of the two study groups is carried out.

Inclusion criteria • Patients with primary knee osteoarthritis set to receive a primary unilateral cemented total knee arthroplasty at Copenhagen University Hospital Hvidovre.

* Participants must be >18 years of age.
* Participants must be able to speak and understand Danish.
* Participants must be able to give informed consent and be cognitively intact.
* Participants must be expected to be able to complete all postoperative controls.
* Participants must not have severe comorbidities, ASA-score ≤ 3. Exclusion criteria
* Terminal illness.
* Rheumatoid arthritis.
* Prior open surgery on the affected knee.
* Prior arthroscopic surgery with surgery on anterior and/or posterior cruciate ligament (meniscal surgery only does not lead to exclusion).
* Prior high-energy trauma to the affected knee.
* Prior history of anterior and/or posterior cruciate ligament rupture.
* Suspicion of anterior and/or posterior cruciate ligament rupture at clinical examination.
* Documented osteoporosis with patient in active medical treatment.
* Comorbidity with altered pain perception (e.g. DM with neuropathy).
* Participants that develop deep infection in the follow-up period are excluded from the study.

Regarding RSA assays

• Participants with less than 3 Tantalum beads visible around the Femur- or Tibia component on RSA assays are excluded from the migration measurements. Data regarding secondary objectives from these subjects will be included.

Regarding intraoperative exclusion • If the anterior and/or posterior cruciate ligaments are found missing or totally ruptured at direct intraoperative visualization, patients excluded at this point and will receive the department's standard prosthesis (Vanguard CR if posterior cruciate ligament is intact).

Regarding contraception

• Patients who receive knee prosthesis have most often reached the non-fertile age (50+). In the case that a fertile woman participates in the study it will be ensured that she is not pregnant.

Intervention group After being allocated to either of the two groups, participants will receive either Vanguard XP or Vanguard CR prosthesis. After discharge outpatient controls are carried out after 3 months, 1, 2, 5, and 10 years postoperatively. RSA assays are performed postoperatively and after 3 months, 1, 2, 5, and 10 years. Patients who meet the inclusion criteria but do not wish to participate in the study will receive the standard treatment for knee osteoarthritis at our institution, which is a cemented TKA and outpatient follow-up 3 months postoperatively.

6. Methods The study is conducted in accordance with the CONSORT statement. The project in 5 steps

1. Project information and signed consent before surgery.
2. Intraoperative assessment of the cruciate ligaments with exclusion of the patient if the anterior and/or posterior cruciate ligaments are found missing or totally ruptured.
3. Surgery with insertion of either Vanguard XP or Vanguard CR prosthesis. Tantalum beads are placed in the bone around the femur- and tibial components. Surgery is performed at Copenhagen University Hospital Hvidovre.
4. Postoperatively, participants are admitted to a dedicated fast track arthroplasty unit and will receive standard treatment after TKA until discharge. Discharge criteria are ability to walk >70 m with crutches or better, ability to get in and out of bed as well as up from a chair, and sufficient oral pain treatment. Before discharge RSA is performed.
5. 3 months and 1, 2, 5. and 10 years postoperatively participants are seen on an outpatient basis.

Demographic data, surgery time and length of hospital stay are also registered.

Surgery procedure Surgery is performed as described in the manufacturer's technical guide. After randomization participants will receive either a cemented Vanguard XP or Vanguard CR prosthesis.

One of three senior surgeons (Henrik Husted, Kristian Otte, Anders Troelsen) dedicated to knee arthroplasty surgery will perform all operations with an assistant.

Technique: A standard medial Para patellar incision is used. Femur and tibial surfaces are prepared using standard cutting guides. When the CR prosthesis is used ACL is resected and PCL is spared. When the XP prosthesis is used both ACL and PCL are spared. The XP prosthesis is used with a tibail tray and a bearing surface for this purpose. A minimum of six 1 mm Tantalum beads are placed in the distal femur and proximal tibia. A sawbones phantom study to detect optimal placement of beads will be performed prior to operation of the first patient. Femur- and tibial components are cemented to the bone. Soft tissue balancing is performed to ensure optimal stability and ROM. An E1-vitamin enriched polyethylene tibial liner is used. Resurfacing of patella is performed in all cases. Joint capsule and subcutis are closed using tied nuts. Skin is closed with staples. No drains are used.

Postoperatively, participants will receive standard pain treatment and rehabilitation until discharge2.

Measurements with RSA Since the 1970ies, RSA has been used to measure the migration of implants in relation to the surrounding bone. Peroperatively, 1 mm Tantalum beads are placed in the bone surrounding the prosthesis using a specialized instrument. Postoperatively, simultaneous radiographs from two different angles are used to visualize distances between the prosthesis and the Tantalum beads three-dimensionally using a special computer software programme (Model Based RSA)3. Then the migration of the prosthesis over time can be calculated. Migration of both the femur- and tibia components can then be calculated.

Radiographs are performed at the Radiological Department, Copenhagen University Hospital Hvidovre. Participants are placed in the supine position and the lower leg is placed on a premade cushion. The x-ray tubes are placed 145 cm above the floor in a mutual angle of 44 degrees (+/-22 degrees relative to the sagittal axis of the participant) so that the path of the beam from each x-ray tube passes through the knee of the participant. Standard x-ray films are placed in a calibration box designed to Model Based RSA. Using Model Based RSA software and pre-scanned models of the prosthesis, the radiographs are used to establish a three-dimensional coordinate presenting the relations between the prosthesis and the Tantalum beads. Distances between the Tantalum beads and the prosthesis can be calculated and subsequently used to calculate migration of the prosthesis over time.

In order to be able to calculate migration of the prosthesis, at least three Tantalum beads around the femur- and tibial components should be visual on the RSA radiographs. If this is not achieved, the participant is excluded from the migration measurements. In order to address this issue at least 6 Tantalum beads are placed in the distal femur and proximal tibia preoperatively.

7. Registrations All registrations are done prospectively. Primary objectives Migration/rotation: Migration of the prosthesis measured by RSA3. Implant-migration/rotation is defined as changes in distances between the prosthesis and the Tantalum beads over time.

Participant perceived knee function: Participant perceived knee function is evaluated preoperatively and at 3 months, 1, 2, 5, and 10 years follow-up using the validated Forgotten Joint Score (FJS)4 and Oxford Knee Score (OKS)5.

Secondary objectives Health related quality of life (HRQoL): Participant perceived HRQoL is evaluated preoperatively and at 3 months, 1, 2, 5, and 10 years follow-up using the validated EQ-5D Range of motion (ROM): Active and passive knee ROM is measured preoperatively and at 3 months, 1, 2, 5, and 10 years follow-up using a goniometer6.

Periprosthetic osteolysis: Radiological signs of periprosthetic osteolysis are evaluated on plain radiographs at 1, 2, 5, and 10 years follow-up.

Knee pain: Knee pain is evaluated at 3 months, 1, 2, 5, and 10 years follow-up using the Visual Analogue Scale (VAS)7 in which 0 represents no pain at all and 10 represents worst pain imaginable.

Satisfaction with the knee: At 3 months, 1, 2, 5, and 10 years participants are asked to describe their satisfaction with the knee using the VAS-scale. 0 is used when the participant is maximally dissatisfied with the knee.

Expectations/fulfilment of expectations: Preoperatively participants are asked about their expectations to the forthcoming knee replacement. At 1, 2, 5, and 10 years follow-up, participants are asked to evaluate how well the knee replacement met their expectations using the VAS-scale. 0 is used when expectations were not fulfilled at all and 10 is used when expectations were fully fulfilled.

Surgery time: Duration from the start of the incision until staples are placed is documented.

Length of hospital stay: Length of hospital stay defined as from the day of surgery until discharge is documented.

Complications: Thrombo-embolic complications, wound healing complications, infections, nerve palsies and revisions are documented.

Peroperative release: If peropertive release (medial, lateral, posterior) is performed in order to obtain stability, this is documented.

8. Risks and adverse effects The risks in this study are related to: 1) Insertion of Tantalum beads in the bone, 2) Additional radiation in relation to the RSA-assays, and 3) The use of a new prosthetic design.

1. Insertion of Tantalum beads in the bone in order to carry out RSA-assays has been done increasingly over the last 25 years. In the literature, no side effects have been reported regarding insertion of Tantalum beads when these have been used for RSA-assays. Tantalum is also used in sutures and staples and has proven bio-convertible and without tendency to corrode bone8-9.
2. In this study RSA-assays are carried out postoperatively and at 3 months, 1, 2, 5, and 10 years follow-up. At 3 months follow-up an additional RSA-assay is performed to ensure the precision of the setup. This means that each participant is exposed to 5 additional RSA-assays. The radiation dose used at each RSA-assay is equivalent to that of conventional radiographs, 0.2 mSV. Each participant is therefore exposed to an additional radiation dose of 1.4 mSV. The background radiation in Denmark is ≈ 2-3 mSV/year. The additional radiation that each participant is exposed to in this study is equivalent to 6-8 months of background radiation. Therefore we believe that the RSA-assays will not cause additional risks for the participants in this study10.
3. In this study a new prosthetic design, the Vanguard XP TKA system (Biomet®, Warsaw, Indiana, USA), is tested. The Vanguard XP system has obtained FDA-approval in the USA and is the further development of the Vanguard system, which has shown good clinical results in earlier studies11-12. We therefore find it highly relevant to investigate the results of primary total knee replacement with the Vanguard XP TKA system. We do not believe that the use of this new prosthetic design will cause additional risks for the participants in this study.

   Investigators Surgery procedures, investigations and radiological assays are carried out by trained medical doctors, nurses, physiotherapists and radiologists associated to the Orthopaedic and Radiology departments at Copenhagen University Hospital Hvidovre.

   Unintended events Unintended events are defined as any unintended and unfavourable occurrences, symptoms or illnesses experienced by the participants in this study, regardless of its coherence with the study.

   Unintended events are documented continuously. Data regarding unintended events will be retrieved from the participant's medical records by the primary investigator. Data from participant medical records will not be disclosed to a third Party.

   Severe unintended events

   Severe unintended events are defined as serious unintended occurrences or side effects that cause:

   • Death.

   • Life threatening situations.

   • Admittance to an intensive care unit.

   • Permanent severe disabilities.

   In the case of a severe unintended event, the investigators of this study are obligated to assess if the event is caused by the interventions introduced in this study, e.g. the insertion of Tantalum beads in the bone. In this assessment, the following factors should be included:
   * Coherence in time.
   * Accordance with known consequences of the treatment or investigations.
   * Alternative reasons for the unintended event. If the severe unintended event is considered caused by the interventions introduced in this study, the project will be terminated ahead of time.

9. Ethics At Copenhagen University Hospital Hvidovre, treatment of osteoarthritis with TKA is mastered on a super-specialist level. We find this study to be highly relevant regarding the potential beneficial effects of the new prosthetic design (Vanguard XP) on postoperative knee function and patient perceived outcome.

The study is conducted in accordance with principals described in the Helsinki declaration.

Participants in the study are covered by the patient insurance of Copenhagen University Hospital Hvidovre.

This protocol, along with written participant information and consent declaration, is to be approved by the local Ethics Committee before enrolments of participants are commenced.

The project will be registered at clinicaltrials.gov. The project will be approved by the Danish Data Protection Agency. It is the responsibility of the primary investigator to inform the local Ethics Committee if any changes are made to the protocol or if any severe adverse effects occur. The primary investigator stores all correspondence regarding the study.

All participants will receive oral and written information about the study before consent. It is the responsibility of the primary investigator that the information to the participant is adequate. Participants are included when signed consent from the participant is obtained. Project information is then given in an undisturbed environment (in a closed examination room) by an authorized investigator of this study. Project information is given at the first outpatient consultation, when treatment with insertion of a TKA is decided. A nurse is present when the information is given. Participants are informed about the right to having a dependent present when project information is given. Participants are informed that a period of consideration of at least 2 weeks is an opportunity along with the right to a second consultation. Signed consent, however, is to be given latest at admittance before surgery.

The oral information is in accordance with the written information and is adjusted to the age, educational level and social conditions of the participant. It is ensured that the participant has understood the content of both the oral and written information before signed consent is given.

It is the responsibility of the primary investigator that the authorized investigator is adequetly informed about the study and academically qualified to giving the oral information.

10. Data recordings Participants in this study are identified with an assigned allocation number. At the end of the study all patient related data are destroyed.

All sensitive personal data regarding participants will be stored in accordance with guidelines presented by the Personal Data Act. Personal data regarding participants will be treated anonymously. The study will be reported to the Danish Data Protection Agency. The primary investigator will process all data. Participants will receive oral and written information concerning the handling of sensitive personal data.

11. Statistics The STATA statistical software will be used when processing data in this study. Comparative statistics will be used based on the distribution of data.

12. Financial conditions This project is financed by Dept. of Orthopaedic Surgery, Copenhagen University Hospital Hvidovre with finantial support from Biomet®, Warsaw, Indiana, USA.

The investigators of this study have independently initiated the project. Besides this study, the primary investigator has no affiliation to Biomet®. 13. Publications The results of this project are expected to be published in an international medical journal. The primary investigator prepares the manuscript, which is approved by the remaining investigators of the project. The results of this study are also expected to be presented at national and international orthopaedic conventions. If publication is not achieved, the results of this study (positive, negative or inconclusive) will be presented on the homepage of our institution.

Co-authorship is awarded according to the Vancouver rules. The investigators will be the authors in the following order:

Morten G. Thomsen, Henrik Husted, Kristian S. Otte, Kasper Gosvig, Anders Troelsen

Biomet will not be able to prevent publication of the results of this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary knee osteoarthritis set to receive a primary unilateral cemented total knee arthroplasty at Copenhagen University Hospital Hvidovre.
* Participants must be >18 years of age.
* Participants must be able to speak and understand Danish.
* Participants must be able to give informed consent and be cognitively intact.
* Participants must be expected to be able to complete all postoperative controls.
* Participants must not have severe comorbidities, ASA-score ≤ 3.

Exclusion Criteria:

* Terminal illness.
* Rheumatoid arthritis.
* Prior open surgery on the affected knee.
* Prior arthroscopic surgery with surgery on anterior and/or posterior cruciate ligament (meniscal surgery only does not lead to exclusion).
* Prior high-energy trauma to the affected knee.
* Prior history of anterior and/or posterior cruciate ligament rupture.
* Suspicion of anterior and/or posterior cruciate ligament rupture at clinical examination.
* Documented osteoporosis with patient in active medical treatment.
* Comorbidity with altered pain perception (e.g. DM with neuropathy).
* Participants that develop deep infection in the follow-up period are excluded from the study.

Regarding RSA assays

• Participants with less than 3 Tantalum beads visible around the Femur- or Tibia component on RSA assays are excluded from the migration measurements. Data regarding secondary objectives from these subjects will be included.

Regarding intraoperative exclusion • If the anterior and/or posterior cruciate ligaments are found missing or totally ruptured at direct intraoperative visualization, patients excluded at this point and will receive the department's standard prosthesis (Vanguard CR if posterior cruciate ligament is intact).

Regarding contraception

• Patients who receive knee prosthesis have most often reached the non-fertile age (50+). In the case that a fertile woman participates in the study it will be ensured that she is not pregnant.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-11; Primary Completion 2017-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
To compare the Vanguard CR and Vanguard XP prosthesis regarding migration/rotation over time, measured by RSA | 2 years
  Migration/rotation of the prosthesis measured in mm/degrees using RSA.

SECONDARY OUTCOMES:
To compare patient reported outcomes after treatment with a Vanguard CR or Vanguard XP prosthesis | 2 years
  Pain (VAS-scale) Satisfaction (VAS-scale) OKS (Oxford knee score) questionnaire FJS (Forgotten Joint Score) questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Orthopedics, University Hospital of Hvidovre, Denmark., Hvidovre, Capital Region of Denmark, Denmark

REFERENCES:
- [Derived] Troelsen A, Ingelsrud LH, Thomsen MG, Muharemovic O, Otte KS, Husted H. Are There Differences in Micromotion on Radiostereometric Analysis Between Bicruciate and Cruciate-retaining Designs in TKA? A Randomized Controlled Trial. Clin Orthop Relat Res. 2020 Sep;478(9):2045-2053. doi: 10.1097/CORR.0000000000001077. PMID 32023233